CLINICAL TRIAL: NCT05579457
Title: Effect of Physical Performance Levels of Elderly Living In Urban and Rural Areas on Social Participation, Social Functioning, and Quality of Life
Brief Title: Physical Performance Levels and Social Participation in Elderly Living In Urban and Rural Areas
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tahir Keskin , Pt, MSc, physical Therapy and Rehabilitation, Suleyman Demirel University
Other Study IDs: 72867572.050.01.04.2953
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Eldrely

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- elderly people living in rural areas
  Interventions: Other: Short Physical Performance Battery
- elderly people living in urban areas
  Interventions: Other: Short Physical Performance Battery

INTERVENTIONS:
Other: Short Physical Performance Battery — The SPPB was applied to determine the physical performance levels of the elderly. This test is a valid and reliable test that measures the performance of the lower extremities and can be applied for elderly. The SPPB included three sections: getting up from a chair, standing balance, and walking speed. At the end of these tests, the scores of the three sections were calculated and higher scores were evaluated as reflecting higher levels of physical performance

SUMMARY:
Purpose: This study aims to investigate the effect of physical performance levels of elderly living in rural and urban areas on social participation, social functioning, and quality of life.

Method: A total of 418 volunteer elderly aged 65 and over living in rural (42.3%) and urban (57.7%) areas participated in this study. The Mini-Mental State Examination, Short Physical Performance Battery, the World Health Organization Quality of Life Scale for Older Adults, Leisure Time subscale of the Social Functioning Scale and the Community Integration Questionnaire were applied to participants.

ELIGIBILITY:
Inclusion Criteria:

* individuals over the age of 65 years who received a score of ≥24 from the Mini-Mental State Examination were included in the study

Exclusion Criteria:

* elderly who were unable to communicate verbally, were unable to move independently, had undergone any operations in the last 6 months, had been diagnosed with cancer, or had severe vision loss, stroke, Parkinson's disease, multiple sclerosis, or other neurological diseases were excluded from the study

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study was carried out with the participation of elderly residing in the provinces of Isparta, Burdur, and Antalya in the Mediterranean region of Turkey
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Community Integration Questionnaire | 02.04.2021
  The questionnaire consists of a total of 18 questions and the highest total score attainable is 35. A total score of 0 is evaluated as no social participation and a total score of 35 is evaluated as full social participation, with an increase in the total score indicating an increase in social participation

SECONDARY OUTCOMES:
Social Functioning Scale ( | 02.04.2021
  The SFS is a tool that evaluates the social role functions of individuals. It has been determined that the SFS is a valid and reliable scale for use in Turkish society

CONTACTS AND LOCATIONS:
Locations (1):
- Tahir KESKİN, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided